CLINICAL TRIAL: NCT00831259
Title: Silent Cerebral Infarcts in Patients With Pulmonary Embolism and a Patent Foramen Ovale: a Prospective Diffusion-weighted Magnetic Resonance Imaging Study.
Brief Title: Risk of Stroke in Pulmonary Embolism With a Patent Foramen Ovale (PFO)
Acronym: ICEP
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Patrick MICHEL, research and strategy manager, CHU de CAEN
Other Study IDs: CHU de Caen
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-05

CONDITIONS: Silent Stroke; Pulmonary Embolism; Patent Foramen Ovale
Keywords: stroke; PFO; embolism
MeSH Terms: conditions — Pulmonary Embolism; Foramen Ovale, Patent; Stroke; Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Incidence of silent stroke in patients with PFO
- 2: Incidence of silent stroke in patients without PFO

SUMMARY:
Pulmonary embolism is associated with a small but definite risk of paradoxical embolism in patients with a patent foramen ovale (PFO). While neurologic complications are unfrequent the incidence of clinically silent brain infarction is unknown. We will assess the rate of clinically apparent and silent cerebral embolism in patients with a pulmonary embolism (PE) in relation to the presence or not of a PFO.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary embolism, informed consent signed, no-contraindication to MRI

Exclusion Criteria:

* contra-indication to MRI, informed consent not obtained

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive series of patients with a pulmonary embolism
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Incidence of cerebral infarcts as detected by Diffusion-weighted MRI | during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- USIC CHU de Caen, Caen, France